CLINICAL TRIAL: NCT07107477
Title: Prospective Randomized Controlled Trial to Evaluate if Tailored Antibiotic and Steroid Therapy Based on the Interleukin-6 (IL-6) Value in Amniotic Fluid Obtained by Amniocentesis in Patients With Premature Rupture of Membranes is Associated With Pregnancy Prolongation Compared to Standard Management.
Brief Title: TAILORED Therapeutic Regime in Patients With Preterm Premature Rupture Of Membranes to Prolong Pregnancy, Improve Maternal and Neonatal Outcomes, and Reduce Antibiotic Burden
Acronym: TAILORED-PROM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Central and Eastern European Gynecologic Oncology Group (Other)
Collaborators: University Hospital Brno (Unknown); General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, David Cibula, Prof. Dr., General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAILORED-PROM 2024-520237-77-0
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Preterm Premature Rupture of Membranes (PPROM)
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes | interventions — Amniocentesis; Neuroprotection; Antibiotic Prophylaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A: TAilored management (Experimental): No steroids at admission Antibiotics - GBS prophylaxis + macrolides always at admission till results of amniotic fluid IL-6 Amniocentesis (Within 24 hours of admission to the hospital)
  * Based on the amniotic fluid IL-6 results:
  * IL-6 ˂ 2600 - discontinuing GBS prophylaxis + macrolides, no steroids.
  * IL-6 ≥ 2600 - Steroids and initial broad spectrum ABX, adjustment according to cultures and PCR
  Interventions: Procedure: Tailored antibiotic and steroid therapy based on the IL-6 value in amniotic fluid obtained by amniocentesis in patients with premature rupture of membranes; Drug: Antenatal steroids administration; Drug: Neuroprotection; Drug: antibiotic prophylaxis
- ARM B: standard care (Active Comparator): Antenatal steroids - always at admission Antibiotics - GBS prophylaxis + macrolides, lasting for 7-10days, then discontinued.
  Interventions: Drug: Antenatal steroids administration; Drug: Neuroprotection; Drug: antibiotic prophylaxis; Drug: Antibiotics administration

INTERVENTIONS:
Procedure: Tailored antibiotic and steroid therapy based on the IL-6 value in amniotic fluid obtained by amniocentesis in patients with premature rupture of membranes — In Arm A, Amniocentesis will be performed once a week until delivery, with a maximum of seven procedures per patient. If the pregnancy continues beyond this period, follow-up will proceed without further amniocentesis.
  * If IL-6 ≥ 2600:
  * steroids and initial broad spectrum ABX will be administered,
  * rotation of ABX according to cultures and PCR.
  * If steroids already administered, a second course can be administered prior to 34+0 if at least 7 days have passed after the previous course.
  Other Names: amniocentesis
  Arms: ARM A: TAilored management
Drug: Antenatal steroids administration — 1. Clinical and/or laboratory signs of chorioamnionitis will result in an intervention consisting of the course of antenatal steroids (if not already administered, or as a single course prior 34+0 if at least 7 days have passed after the previous course), initial broad spectrum antibiotics, or delivery, depending on the week of pregnancy and clinical status.
  2. Uterine activity with progression of vaginal finding will result in course of antenatal steroids (if not already administered, or as a single course prior 34+0 if at least 7 days have passed after the previous course) and tocolysis
Drug: Neuroprotection — In patients with imminent preterm birth prior 32+0 week of pregnancy, foetal neuroprotection will be administered consisting of MgSO4 in an intravenous loading dose of 4 g (administered slowly over 20-30 min), followed by a 1 g per hour maintenance dose. This regimen should continue until birth but should be stopped after 24 h if undelivered.
Drug: antibiotic prophylaxis — Antibiotics - Group B Streptococcus (GBS) prophylaxis + macrolides, always at admission.
Drug: Antibiotics administration — 1. GBS prophylaxis + macrolides: Penicillin G (benzylpenicillin) 5mil IU IV initially and then 2-3 IU (dose adjusted to body weight) IV every 4h twice, then every 6h + Clarithromycin 500mg po every 12h for 7-10 days or till delivery.
  2. Initial broad spectrum ABX: Ampicillin/sulbactam 3g IV every 6 hours + Gentamicin 5 mg/kg IV (<60 kg 240 mg, 61-80 kg 320 mg, >80 kg 400 mg) every 24h for 5-7 days according to the clinical state.
  Comments:
  Alternative ABX in patients with allergy to PCN/AMP: Vancomycin 1g IV every 12 h or Clindamycin 600-900g IV every 8h taking antibiotic sensitivity into account.
  Before administering the third dose of gentamicin, its serum level should be determined (at a level >4 umol/l, the dose must be reduced).
  Arms: ARM B: standard care

SUMMARY:
The goal of this clinical trial is to learn whether tailoring antibiotic and steroid treatment based on a lab result (interleukin-6, or IL-6) from amniotic fluid can help safely prolong pregnancy in people with preterm premature rupture of membranes (pPROM). This condition means the water breaks too early, before 37 weeks of pregnancy, which increases the risk of infection and early birth.

The main questions the study aims to answer are:

1. Can using IL-6 levels to guide treatment help the pregnancy last more than 7 days after pPROM?
2. Can this approach improve health outcomes for both the parent and the baby?

Researchers will compare two groups:

1. A tailored treatment group, where IL-6 levels from amniotic fluid help decide when to give steroids and antibiotics.
2. A standard care group, where everyone receives the same treatment right after diagnosis.

Participants will:

* Be screened to confirm pPROM and eligibility.
* Be randomly assigned to one of the two groups.
* Receive regular check-ups and monitoring in the hospital until delivery.
* In the tailored group, have weekly amniocentesis (a safe procedure to collect amniotic fluid) if needed.

The study includes follow-up for 6 months after birth to track both the baby's and parent's health.

This research may help doctors better time treatments, reduce unnecessary use of medications, and improve outcomes for families facing pPROM.

ELIGIBILITY:
Inclusion Criteria:

* pPPROM Confirmed by Amnisure test1 and/or clinical signs of pPROM on examination (Clinical signs of pPROM: presence of visual pooling of amniotic fluid during sterile speculum examination)
* Weeks of pregnancy 22+03 - 33+64
* Singleton pregnancy
* Signed informed consent form (ICF)
* Completely uncomplicated pregnancy until the occurrence of pPROM

Exclusion Criteria:

* active labour (uterine activity leading to cervical dilatation greater than 4 cm)
* Obstetrical reason for immediate delivery such as heavy vaginal bleeding, prolapsed cord, or foetal distress
* Multiple pregnancy
* Pregnancy with chromosomal or severe morphological abnormality
* Signs of chorioamnionitis at the admission (clinical and/or laboratory)
* Patients with severe immunological compromise (immunodeficient)
* Patients with an oncological disease/immunosuppression
* Patients with an active drug abuse
* Non-compliant patients
* Any contraindication according to the valid SmPC for the administered product

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
The latency of pregnancy of more than 7 days from premature rupture of membranes to delivery | From enrollment to the delivery (0-98 days).
  Latency ˃ 7d is an outcome traditionally used in trials studying pPROM and PTB.

SECONDARY OUTCOMES:
Latency to birth | Measured in days from pPROM to birth (0-98 days).
Incidence of chorioamnionitis and funisitis | From the enrollment to the delivery (0-98 days).
  Diagnosed during pregnancy based on clinical criteria or postpartum based on histological examination of placenta and umbilical cord.
Short-term adverse maternal outcomes | From the enrollment to the 6 weeks postpartum. Time from enrollment to delivery is 0-14 weeks. Time frame ranges from 0-20 weeks.
  List of short-term adverse maternal outcomes:
  1. mortality
  2. infection complication: sepsis, endometritis, wound infection, endometritis
  3. postpartum haemorrhage
  4. postpartum hysterectomy
  5. admission to the maternal intensive care unit
  6. unplanned operative procedure after delivery (dilation and curettage, laparoscopy, or laparotomy)
  7. injury requiring repair
  8. uterine rupture
  9. haemorrhage of >1000 mL
  10. transfusion
  11. acute renal insufficiency
  12. venous thromboembolism
  13. pulmonary embolism
  14. readmission to the hospital within 6 weeks
Short-term neonatal outcomes | From the birth to 6-months postpartum.
  List of short-term neonatal outcomes:
  1. mortality
  2. gestational week at birth, birth weight and weight percentile
  3. status of antenatal steroids (expired/complete/incomplete)
  4. umbilical cord pH
  5. IL-6 from the umbilical cord
  6. Apgar score at 1 and 5 minutes
  7. need of intubation of the neonate after birth
  8. surfactant application
  9. days on ventilator
  10. the length of non-invasive respiratory support (postmenstrual week)
  11. the need for home oxygen therapy
  12. early pulmonary hypertension with iNO (Inhaled nitric oxide)
  13. patent ductus arteriosus (PDA) over 14 days over 1.5 mm/ ligation/ left ventricular outflow (LVO) over 450 ml/kg/min in 14 days)
  14. intraventricular haemorrhage (IVH) stage III-IV or periventricular leukomalacia (PVL) or other severe injury of brain visible on ultrasound
  15. bronchopulmonary dysplasia (BPD) stage II and III (Jensen)
  16. retinopathy of newborn (ROP) requiring invasive treatment
  17. necrotizing enterocolitis (NEC) with need of surgical so

OTHER OUTCOMES:
Microbiome in mother and newborn | Samples collected immediatelly after delivery.
  Microbiome sequencing based on the bucal and rectal swabs.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - University Hospital Brno, Brno
  - General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: Undecided
Only IPD used in the results publication

REFERENCES:
- [Background] Obrich E. Telephone reassurance program's first year. Home Healthc Nurse. 1998 Jan;16(1):11-2. doi: 10.1097/00004045-199801000-00002. No abstract available. PMID 9469066
- [Background] Filippi M, Campi A, Dousset V, Baratti C, Martinelli V, Canal N, Scotti G, Comi G. A magnetization transfer imaging study of normal-appearing white matter in multiple sclerosis. Neurology. 1995 Mar;45(3 Pt 1):478-82. doi: 10.1212/wnl.45.3.478. PMID 7898700
- [Background] Daum KM, Hill RM. Human tears: glucose instabilities. Acta Ophthalmol (Copenh). 1984 Jun;62(3):472-8. doi: 10.1111/j.1755-3768.1984.tb08427.x. PMID 6464692
- [Background] Ito J, Taura A, Fujita S, Ishiko T, Ishikawa K. Use of rotation flap in the treatment of cutaneous ulceration after cochlear implantation. Otolaryngol Head Neck Surg. 1999 Dec;121(6):830-2. doi: 10.1053/hn.1999.v121.a94251. No abstract available. PMID 10580248
- [Background] Nielsen VG, Andersen JB. [Acid secretion in patients with duodenal ulcer. Comparison of medical and surgical patients]. Ugeskr Laeger. 1970 Dec 3;132(49):2337-40. No abstract available. Danish. PMID 5488235
- [Background] Martins E Silva J. [Perspectives and clinical importance of hemorrheology--influence of erythrocyte deformability]. Acta Med Port. 1984 Apr-May;5(4-5):151-3. No abstract available. Portuguese. PMID 6464808
- [Background] Jen YM, Hendry JH. The distribution of colony-forming cells in the kidney. Cell Prolif. 1993 May;26(3):263-9. doi: 10.1111/j.1365-2184.1993.tb00024.x. PMID 8324073
- [Background] Jammet H, Dousset M. [Role of 2 international agencies (U.S.C.E.A.R. and I.C.R.P.) in radiologic protection]. Rev Epidemiol Sante Publique. 1982;30(2):265-73. No abstract available. French. PMID 7134569
- [Background] Hurme M. Both interleukin 1 and tumor necrosis factor enhance thymocyte proliferation. Eur J Immunol. 1988 Aug;18(8):1303-6. doi: 10.1002/eji.1830180824. PMID 3262066
- [Background] Goodrich JA, Sylvester R. Marketing EAPs: issues and prospects. J Ambul Care Mark. 1992;5(1):197-207. No abstract available. PMID 10122752
- [Background] Boettcher LB, Clark EAS. Neonatal and Childhood Outcomes Following Preterm Premature Rupture of Membranes. Obstet Gynecol Clin North Am. 2020 Dec;47(4):671-680. doi: 10.1016/j.ogc.2020.09.001. Epub 2020 Oct 7. PMID 33121652
- [Background] Prelabor Rupture of Membranes: ACOG Practice Bulletin, Number 217. Obstet Gynecol. 2020 Mar;135(3):e80-e97. doi: 10.1097/AOG.0000000000003700. PMID 32080050